CLINICAL TRIAL: NCT04376437
Title: The Kinetics of Endocannabinoids in Patients With Chemotherapy Induced Peripheral Neuropathy by Using a Portable Metered-Dose Cannabis Inhaler
Brief Title: The Kinetics of Endocannabinoids in Patients With Chemotherapy Induced Peripheral Neuropathy by Using Medical Cannabis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Syqe Medical (Industry)
Responsible Party: Principal Investigator, Gil Bar Sela, Oncologist, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ENDO-CIPN 1
Record Dates: First submitted 2019-10-31; First posted 2020-05-06 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Medical Marijuana

STUDY DESIGN:
Intervention Model Description: Syqe Medical Cannabis inhaler is approval medical device in Israel , this is only Basic science study with main purpose to learn more about the kinetics of endocannabinoids .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- medical cannabis (Experimental): All patients will start with 250mcg cannabis flos BID and will follow the titration plan of dose modification according to CIPN relief and adverse events. Maximum dose of 2,000mcg per day is prescribed at the end of titration period, which is continuous for 15 days (about 2 weeks).On 10 weeks visit all patients will be discontinued from the treatment. In case of worsening of neuropathy at any point during the 4 weeks of FU, patients might be able to restart with inhaled MC treatment for no more than 4 weeks. Total treatment in this study will be for no more than 14 weeks.
  Interventions: Drug: medical cannabis

INTERVENTIONS:
Drug: medical cannabis — inhalation by using a Portable Metered-Dose Cannabis Inhaler
  Other Names: medical marijuana

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is the most common neurological cancer treatment complication. Medical cannabis is indicated in Israel for the treatment of chronic pain, spasticity and for the control of pain and other symptoms in patients with cancer.

The proposed study aims are to study about the changes in level of endocannabinoids following continuous exposure to phytocannabinoids and about the long-term effect of medical cannabis on CIPN.

DETAILED DESCRIPTION:
This will be a self-titrated, open-label design study. Subjects who begin taxanes or oxaliplatine therapy and were diagnosed with CIPN will be recruited to the study.

After providing their written informed consent, the study physician obtained a medical history, demographic details and conducted a physical examination. During the current study, baseline period for CIPN evaluation will be 2 weeks, while patients will fill several questionnaires. Baseline CIPN will be evaluating by DN4 and BPI questionnaires. EQ-5D and PSQI will be filled for baseline Quality of life (QOL) and sleepiness status, accordingly.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age above 18 years and below 80 years old. 2. Pathology of Breast or GI malignancies. 3. Treatment with Taxans (Taxol/ Taxotere) or Oxaliplatin for adjuvant treatment or metastatic disease.

  4. Estimated life expectancy ≥ 6 months. 5. Performance status ≤1 (ECOG classification). 6. Sign of written informed consent. 7. CIPN is examined during the chemotherapy treatment DN4 score must be above 4 (and by physician decision) for more than one week.

  8. Patient with adequate liver/renal function at screening as described:
  * Creatinine clearance >30 ml/min as calculated by Cockcroft-Gault Equation.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN. 9. Patients who suffer from pain although using a stable analgesic treatment' at least 14 days before entering the trial (no limitation for the use of the analgesic).

    10. Patient possessed a valid license from the Israeli Ministry of Health to receive medicinal cannabis.

    11. Patient is able and willing to comply with study requirements. 12. Patient agrees to use only medical cannabis provided by study team until the end of study period.

    13. Patient has not undergone major surgery in the month prior to the study start.

    14. Patient agrees not to participate in other interventional clinical trial during the study participation.

Exclusion Criteria:

* 1. Use of cannabis or synthetic cannabinoids in the last two weeks (urine test for cannabinoids are positive).

  2. Patient with known or past substance abuse. 3. Patients with major psychiatric disorders (e.g. schizophrenia, dementia, and intellectual disabilities).

  4. Patients with first degree siblings under the age of 30 years old with psychiatric disorders.

  5. Patients with uncontrolled diabetes mellitus, cardiovascular, or convulsive disorders according to investigator.

  6. Patients with sensitivity to cannabis or cannabinoids. 7. Patients with known neuropathic pain due to diabetes or other diseases. 8. Patients with severe respiratory disease. 9. Patients with brain metastases or brain tumors may participate if completed radiotherapy treatment at least 14 days prior to signing the informed consent and last imaging did not show any worsening.

  10. Female subjects who are pregnant, lactating, or want to get pregnant during the study period and one month following the study. Male subjects who want their partner to get pregnant during the study period and one month following the study.

  11. Females of childbearing potential or males whose partners with childbearing potential and did not use adequate contraceptives 28 days prior to study start or during the study.

  12. Other life-threatening medical conditions that disqualify the patient from participating in the study, according to the Primary Investigator's judgment.

  13. Anticipated alcohol or barbiturate use during the study period. 14. Participation in other clinical trials during the last month. 15. Subjects who are using one of the following medications: opiates (Primidone, Phenobarbitol, Arbamazepine, Rifampicin, Rifabutin, Troglitazone and Hypericum perforatum).

  16. Patient who has undergone a major surgery a month prior to study start.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the level of 150 different endocannabinoids. | Determined on blood samples collected during the 4 months of participation in the study
  Circulating endocannabinoids concentrations .

SECONDARY OUTCOMES:
Changes from the baseline of neuropathic pain during medical cannabis treatment . | during 4 months of participation in the study
  Neuropathic pain detected by DN4 questionnaire .
Changes in Quality of life by FACT-GOG-Ntx | This exam will be performed every visit.during 4 months of participation in the study
  Changes of Quality of life will be evaluated by Functional Assessment of Cancer Therapy - Gynecologic Oncology Group-Neurotoxicity ( FACT-GOG-Ntx) questionnaire
Changes in Quality of life by BPI | This exam will be performed every visit.during 4 months of participation in the study
  Changes of Quality of life will be evaluated by BRIEF PAIN INVENTORY (BPI) tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek MC, Afula, North, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pachman DR, Watson JC, Loprinzi CL. Therapeutic strategies for cancer treatment related peripheral neuropathies. Curr Treat Options Oncol. 2014 Dec;15(4):567-80. doi: 10.1007/s11864-014-0303-7. PMID 25119581
- [Result] Hammack JE, Michalak JC, Loprinzi CL, Sloan JA, Novotny PJ, Soori GS, Tirona MT, Rowland KM Jr, Stella PJ, Johnson JA. Phase III evaluation of nortriptyline for alleviation of symptoms of cis-platinum-induced peripheral neuropathy. Pain. 2002 Jul;98(1-2):195-203. doi: 10.1016/s0304-3959(02)00047-7. PMID 12098632
- [Result] Mitchell PL, Goldstein D, Michael M, Beale P, Friedlander M, Zalcberg J, White S, Thomson JA, Clarke S. Addition of gabapentin to a modified FOLFOX regimen does not reduce oxaliplatin-induced neurotoxicity. Clin Colorectal Cancer. 2006 Jul;6(2):146-51. doi: 10.3816/CCC.2006.n.032. PMID 16945171
- [Result] Rao RD, Flynn PJ, Sloan JA, Wong GY, Novotny P, Johnson DB, Gross HM, Renno SI, Nashawaty M, Loprinzi CL. Efficacy of lamotrigine in the management of chemotherapy-induced peripheral neuropathy: a phase 3 randomized, double-blind, placebo-controlled trial, N01C3. Cancer. 2008 Jun 15;112(12):2802-8. doi: 10.1002/cncr.23482. PMID 18428211
- [Result] Abrams DI, Jay CA, Shade SB, Vizoso H, Reda H, Press S, Kelly ME, Rowbotham MC, Petersen KL. Cannabis in painful HIV-associated sensory neuropathy: a randomized placebo-controlled trial. Neurology. 2007 Feb 13;68(7):515-21. doi: 10.1212/01.wnl.0000253187.66183.9c. PMID 17296917
- [Result] Ellis RJ, Toperoff W, Vaida F, van den Brande G, Gonzales J, Gouaux B, Bentley H, Atkinson JH. Smoked medicinal cannabis for neuropathic pain in HIV: a randomized, crossover clinical trial. Neuropsychopharmacology. 2009 Feb;34(3):672-80. doi: 10.1038/npp.2008.120. Epub 2008 Aug 6. PMID 18688212
- [Result] Ware MA, Wang T, Shapiro S, Robinson A, Ducruet T, Huynh T, Gamsa A, Bennett GJ, Collet JP. Smoked cannabis for chronic neuropathic pain: a randomized controlled trial. CMAJ. 2010 Oct 5;182(14):E694-701. doi: 10.1503/cmaj.091414. Epub 2010 Aug 30. PMID 20805210
- [Result] Andreae MH, Carter GM, Shaparin N, Suslov K, Ellis RJ, Ware MA, Abrams DI, Prasad H, Wilsey B, Indyk D, Johnson M, Sacks HS. Inhaled Cannabis for Chronic Neuropathic Pain: A Meta-analysis of Individual Patient Data. J Pain. 2015 Dec;16(12):1221-1232. doi: 10.1016/j.jpain.2015.07.009. Epub 2015 Sep 9. PMID 26362106
- [Result] Boychuk DG, Goddard G, Mauro G, Orellana MF. The effectiveness of cannabinoids in the management of chronic nonmalignant neuropathic pain: a systematic review. J Oral Facial Pain Headache. 2015 Winter;29(1):7-14. doi: 10.11607/ofph.1274. PMID 25635955
- [Result] Lynch ME, Campbell F. Cannabinoids for treatment of chronic non-cancer pain; a systematic review of randomized trials. Br J Clin Pharmacol. 2011 Nov;72(5):735-44. doi: 10.1111/j.1365-2125.2011.03970.x. PMID 21426373
- [Result] Pascual D, Goicoechea C, Suardiaz M, Martin MI. A cannabinoid agonist, WIN 55,212-2, reduces neuropathic nociception induced by paclitaxel in rats. Pain. 2005 Nov;118(1-2):23-34. doi: 10.1016/j.pain.2005.07.008. Epub 2005 Oct 4. PMID 16213089
- [Result] Rahn EJ, Makriyannis A, Hohmann AG. Activation of cannabinoid CB1 and CB2 receptors suppresses neuropathic nociception evoked by the chemotherapeutic agent vincristine in rats. Br J Pharmacol. 2007 Nov;152(5):765-77. doi: 10.1038/sj.bjp.0707333. Epub 2007 Jun 18. PMID 17572696
- [Result] Grotenhermen F. Pharmacokinetics and pharmacodynamics of cannabinoids. Clin Pharmacokinet. 2003;42(4):327-60. doi: 10.2165/00003088-200342040-00003. PMID 12648025
- [Result] Eisenberg E, Ogintz M, Almog S. The pharmacokinetics, efficacy, safety, and ease of use of a novel portable metered-dose cannabis inhaler in patients with chronic neuropathic pain: a phase 1a study. J Pain Palliat Care Pharmacother. 2014 Sep;28(3):216-25. doi: 10.3109/15360288.2014.941130. Epub 2014 Aug 13. PMID 25118789
- [Result] Zusman SP, Lustig JP, Bin Nun G. Cost evaluation of two methods of post tooth extraction hemostasis in patients on anticoagulant therapy. Community Dent Health. 1993 Jun;10(2):167-73. PMID 8402303
- [Result] Skrabek RQ, Galimova L, Ethans K, Perry D. Nabilone for the treatment of pain in fibromyalgia. J Pain. 2008 Feb;9(2):164-73. doi: 10.1016/j.jpain.2007.09.002. Epub 2007 Nov 5. PMID 17974490
- [Result] La Porta C, Bura SA, Llorente-Onaindia J, Pastor A, Navarrete F, Garcia-Gutierrez MS, De la Torre R, Manzanares J, Monfort J, Maldonado R. Role of the endocannabinoid system in the emotional manifestations of osteoarthritis pain. Pain. 2015 Oct;156(10):2001-2012. doi: 10.1097/j.pain.0000000000000260. PMID 26067584
- [Result] Jhaveri MD, Sagar DR, Elmes SJ, Kendall DA, Chapman V. Cannabinoid CB2 receptor-mediated anti-nociception in models of acute and chronic pain. Mol Neurobiol. 2007 Aug;36(1):26-35. doi: 10.1007/s12035-007-8007-7. Epub 2007 Oct 2. PMID 17952647
- [Result] Berman P, Futoran K, Lewitus GM, Mukha D, Benami M, Shlomi T, Meiri D. A new ESI-LC/MS approach for comprehensive metabolic profiling of phytocannabinoids in Cannabis. Sci Rep. 2018 Sep 24;8(1):14280. doi: 10.1038/s41598-018-32651-4. PMID 30250104
- [Result] Vulfsons S, Ognitz M, Bar-Sela G, Raz-Pasteur A, Eisenberg E. Cannabis treatment in hospitalized patients using the SYQE inhaler: Results of a pilot open-label study. Palliat Support Care. 2020 Feb;18(1):12-17. doi: 10.1017/S147895151900021X. PMID 31196236